CLINICAL TRIAL: NCT00436241
Title: A Open Label Study of the Effect of First-line Therapy With Xeloda in Combination With Oxaliplatin on Overall Response Rate in Patients With Locally Advanced and/or Metastatic Gastric Cancer
Brief Title: A Study of Xeloda (Capecitabine) as First-Line Chemotherapy in Patients With Advanced or Metastatic Gastric Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20734
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: Oxaliplatin — 85mg/m2 iv on day 1 of each 2 week cycle
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-10 of each 2 week cycle

SUMMARY:
This single arm study will assess the efficacy and safety of Xeloda in combination with oxaliplatin as first-line chemotherapy in patients with advanced and/or metastatic gastric cancer who have had no prior chemotherapy for advanced or metastatic disease. Eligible patients will receive Xeloda 1000mg/m2 po twice daily, D1-D10 every 2 weeks (10 days treatment followed by 4 days rest period) plus oxaliplatin 85 mg/m2/day iv, D1 every 2 weeks. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* gastric cancer with unresectable locally advanced and/or metastatic disease;
* >=1 measurable lesion;
* ambulatory, with ECOG Performance Status >=1.

Exclusion Criteria:

* previous chemotherapy (except adjuvant or neoadjuvant treatment >=6 months prior to enrollment);
* clinically significant cardiac disease or myocardial infarction within last 12 months;
* CNS metastases;
* history of other malignancy within last 5 years, except for cured basal cell cancer of the skin, or in situ cancer of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Event driven

SECONDARY OUTCOMES:
Time to disease progression, overall survival, duration of response, time to response. | Event driven
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Taiwan (8):
  - Chai Yi
  - Kaohsiung City
  - Keelung
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
  - Yilan